CLINICAL TRIAL: NCT03371186
Title: Implementing an Integrated RMNCH Intervention by Community Health Workers in Achham and Dolakha: National Pilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Possible (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); Ministry of Health and Population, Nepal (Other Government); Planned Parenthood League of Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RMNCHnyaya; 1DP5OD019894-01 (NIH); AID-OAA-A-11-0001 (Other Grant/Funding Number: United States Agency for International Development)
Record Dates: First submitted 2017-12-04; First posted 2017-12-13 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Reproductive, Maternal, Newborn, and Child Health; Integrated, Community-Health Systems
Keywords: Implementation Research; Maternal Mortality and Morbidity; Neonatal Mortality and Morbidity; Infant Mortality and Morbidity; Child Mortality and Morbidity; Community Health Workers; Health Systems Strengthening
MeSH Terms: conditions — Maternal Death; Infant Death | interventions — Community Health Workers; Postnatal Care

STUDY DESIGN:
Intervention Model Description: Stepped wedge, cluster-controlled implementation science trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bundled RMNCH Intervention (Experimental): Stepped wedge, cluster-controlled implementation science trial of 5 bundled intervention components (1. Community Health Worker, 2, Continuous Surveillance, 3. CB-Integrated Management of Newborn and Childhood Illness, 4. Group Antenatal and Postnatal Care, and 5. Balanced Post-Partum Contraceptive Counseling) implemented across 40 village clusters in Achham District, Nepal and 40 village clusters in Dolakha District, Nepal (covering a total population of approximately 300,000) in coordination with district authorities and study staff. The investigators anticipate the experimental arm will enroll approximately 12,000 women and their children over the 18mo enrollment period.
  Interventions: Other: Community Health Worker; Other: Continuous Surveillance; Other: CB-Integrated Management of Newborn and Childhood Illness; Other: Group Antenatal and Postnatal Care; Other: Balanced Post-Partum Contraceptive Counseling

INTERVENTIONS:
Other: Community Health Worker — The intervention is designed to address these primary drivers of underutilization of reproductive, maternal, newborn, and child health services in rural Nepal, namely: poverty, lack of social support, and poor birth planning. The investigators have worked with a cadre of Community Healthcare Workers who, in addition to the responsibilities of local community health volunteers, have added responsibilities, training, and managerial support. These women support their community members in their homes to identify and overcome social barriers and plan for emergency healthcare needs. The goals are to increase utilization of services, maternal and neonatal health knowledge, self-efficacy, social support, and emergency planning among mothers
Other: Continuous Surveillance — Each patient identified by a Community Health Worker will undergo a complete diagnostic evaluation by the hospital-based clinicians and will be enrolled in the study only if they are identified as currently pregnant, have recently given birth, or have a child under the age of 24 months. Continuous surveillance systems ensure that the entire population is surveyed every three months and has a three month touchpoint with a Community Health Worker.
Other: CB-Integrated Management of Newborn and Childhood Illness — Safe delivery care; effective neonatal resuscitation; management of childhood diarrhea, malnutrition, and pneumonia; and treatment of traumatic and congenital surgical conditions can reduce child mortality. Community Based Integrated Management of Newborn and Child Illness (CB-IMNCI) has shown substantial reductions in neonatal and early child mortality. Community Health Workers will use CB-IMNCI as the clinical protocol for ongoing care to the community.
Other: Group Antenatal and Postnatal Care — The proposed model will change antenatal and pediatric care in three major ways: 1) conduct care in a group setting, 2) provide expert and facilitated peer counseling, and 3) incorporate emergency planning. The group setting is designed to create a supportive social network among women facing similar challenges. The opportunity for counseling beyond the current standard will promote detailed emergency planning and the sharing of context-specific advice from peers to overcome barriers to access care. This intervention draws on the strength within communities of women to change health-seeking behaviors.
Other: Balanced Post-Partum Contraceptive Counseling — Research on interventions to improve postpartum contraception suggest strategies that bridge the continuum of reproductive health care-antenatal care, labor and delivery, postnatal care, and infant care-are more effective than short term, stand-alone counseling sessions. The structured counseling module incorporated in the intervention will be partially adapted from the Balanced Counseling Strategy, an interactive contraceptive counseling method developed by the Population Council in accordance with the World Health Organization's tiered effectiveness guidelines. Prior studies in clinical settings in Nepal have demonstrated increased uptake of modern contraceptive methods, especially of long-acting reversible contraceptives with use of balanced counseling.

SUMMARY:
The investigators will conduct a cluster-controlled, stepped wedge implementation science trial of a bundled reproductive, maternal, neonatal, and child healthcare (RMNCH) delivery intervention within an approximate population of 300,000 people in rural Nepal. This intervention integrates five evidence-based approaches for reproductive, maternal, newborn, and child health focused on the "golden 1000 days" from conception through age two: 1) Community Health Worker model of home-based care to monitor and increase utilization of services, maternal and neonatal health knowledge, self-efficacy, social support, and emergency planning among mothers; 2) Continuous surveillance of all pregnancies and children via an integrated electronic medical record; 3) Delivering community-based integrated management of newborn and childhood illness (CB-IMNCI) via CHWs; 4) Group antenatal and postnatal care to improve care delivery and reduce mortality during the "golden 1000 days" from conception to age two; and 5) Balanced counseling to increase post-partum contraception.

ELIGIBILITY:
Inclusion Criteria:

1. Reproductive aged women 15-49;
2. Reproductive aged women 15-49; recently delivered in past two years;
3. Reproductive aged women 15-49; active pregnancy during study period and identified by a CHW serving their village
4. Children aged 0-2; children of recently-delivered mothers (population #2 or #3 above);
5. Healthcare staff; CHWs serving village clusters, CHW Leaders serving one of the village clusters, Nyaya Health Nepal and Government of Nepal employees involved in study design, program implementation, data collection, or data analysis processes; and
6. Must reside in either Achham or Dolakha District, Nepal.

Exclusion Criteria:

Patients meeting inclusion criteria and consenting to study enrollment, as stated above, will be included in the study unless 1) patients migrate from the study are before completion of any of the bundled interventions; 2) patients request exclusion from the study at any point during the bundled intervention.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12000 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Institutional Birth Rate | 3 years
  The percentage of births in a healthcare facility with a healthcare professional present.
Under-Two Mortality Rate | 3 years
  The under-2 mortality rate is the probability (expressed as a rate per 1,000 live births) of a child born in a specified year dying before reaching the age of two if subject to current age-specific mortality rates.
Post-Partum Contraceptive Prevalence Rate | 3 years
  The post-partum contraceptive prevalence rate is number of married reproductive aged women (15-49) in the study population who delivered in the past two years who are using a modern contraceptive method out of the total number of married reproductive aged women (15-49) in the study population who delivered in the past two years.

SECONDARY OUTCOMES:
Home Visit Coverage | 3 months
  The percentage of children under 2 receiving monthly home based care by a CHW out of total number of children under 2 (aggregated by the percentage of pregnant women and reproductive-aged women).
Group Care Content Fidelity | 3 months
  The percentage of topics covered and completed out of total planned topics
Group Participation | 3 months
  The percentage of participants completing group sessions out of total scheduled participants
Session Completion | 3 months
  The percentage of group sessions completed out of total appropriate number of group sessions
First-Trimester Pregnancies Identified | 3 months
  The percentage of pregnancies identified at less than 12 weeks
Antenatal Care Completion | 3 months
  The percentage of women who have had 4 or more antenatal care visits and are eligible for the government financial incentive out of total number of women delivered
Pediatric Pneumonia Incidence | 1 month
  The number of new cases of pneumonia in catchment area in children under age of two/month
Pediatric Diarrhea Incidence | 1 month
  The number of new cases of diarrhea in catchment area in children under age of two/month
Pediatric Stunting Prevalence | 1 month
  The number of cases children in catchment area under age of two whose length-for height or height-for-age is two SDs below WHO Child Growth Standards median/total number of children in catchment area under age of two
Exclusive Breastfeeding Prevalence | 1 month
  The number of infants in catchment area age zero-five months who are exclusively breastfed/total infants in catchment area age zero-five months
Percent of postpartum women with unmet need for contraception | 3 years
  The number of reproductive age women within the first year following the birth of their most recent child who desire to either stop or postpone childbearing for the next 2 years who are not currently using a contraceptive method or have a repeat unintended pregnancy while not using contraception/Total number of women who are up to one year postpartum, excluding women who declare that they are infecund, have had a hysterectomy, or are in menopause
Contraceptive Method Mix | 3 months
  The percentage of women using each method of modern contraception out of total number of women using modern contraception
Total Intervention Cost | 3 years
  The total sum costs of each intervention component
Cost-Effectiveness of Bundled Intervention | 3 years
  The total sum costs of each intervention component over under-2 deaths averted by intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sheela Maru, MD, MPH, Principal Investigator — Possible; Pushpa Chaudhari, MD, Principal Investigator — Ministry of Health and Population, Nepal
Locations (2):
- Nepal (2):
  - Bayalpata Hospital, Sanfebagar, Achham
  - Charikot Primary Health Center, Bhimeshwor, Dolakha

REFERENCES:
- [Derived] Maru S, Nirola I, Thapa A, Thapa P, Kunwar L, Wu WJ, Halliday S, Citrin D, Schwarz R, Basnett I, Kc N, Karki K, Chaudhari P, Maru D. An integrated community health worker intervention in rural Nepal: a type 2 hybrid effectiveness-implementation study protocol. Implement Sci. 2018 Mar 29;13(1):53. doi: 10.1186/s13012-018-0741-x. PMID 29598824